CLINICAL TRIAL: NCT02891512
Title: Effectiveness of Very Low Frequency Magnetic Fields Versus the Supplement "Xinepa" in the Treatment of the Carpal Tunnel Syndrome: Randomized Double-blind Controlled Clinical Trial.
Brief Title: Very Low Frequency Magnetic Fields Versus the Supplement "Xinepa" in the Treatment of the Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, Medical Director, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2545/15
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Magnetic Fields; Pain; Paresthesia; Visual Analogue Scale
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain; Paresthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ELF and Xinepa® (Experimental): The very low frequency magnetic fields (ELF) are magnetic fields already use for orthopedics pathology that have shown to be able to repair, to reduce pain, inflammation and edema in the damaged tissues. Xinepa® is a dietary supplement containing alpha-lipoic acid, N-acetyl-L-carnitine, turmeric, vitamins B, E and C. They have an antioxidant and anti-inflammatory action on nervous system and they act on cellular energy metabolism.
  Interventions: Other: ELF; Other: Xinepa®
- ELF and Placebo Xinepa® (Placebo Comparator): The very low frequency magnetic fields (ELF) are magnetic fields already use for orthopedics pathology that have shown to be able to repair, to reduce pain, inflammation and edema in the damaged tissues. Xinepa® without its specific activity for the condition being treated.
  Interventions: Other: ELF; Other: Placebo Xinepa®

INTERVENTIONS:
Other: ELF — Very low frequency magnetic fields (ELF) at intensity of 100 mT and a frequency of 1-80 Hz. Protocol (antiedema-antinflammatory): 12 sessions, 3 times a week for 4 consecutive weeks, each session lasted 30 minutes.
Other: Xinepa® — 2 tablets of Xinepa daily (morning and evening) for 1 month.
  Arms: ELF and Xinepa®
Other: Placebo Xinepa® — 2 tablets of Xinepa placebo daily (morning and evening) for 1 month.
  Arms: ELF and Placebo Xinepa®

SUMMARY:
The purpose of the study is to determine the effectiveness of the treatment with very low frequency magnetic fields (ELF) on the reduction of pain and the relief of the associated signs such as sensitivity disorders that affect the first three fingers and half of the fourth finger of the hand in patients with carpal tunnel syndrome versus the supplement (= Xinepa).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of carpal tunnel syndrome

Exclusion Criteria:

* Pregnancy;
* Pacemaker or other metallic implants;
* Systemic infectious disorders;
* Neoplastic disorders;
* Epilepsy;
* Severe heart disease.
* Known hypersensitivity to the components of Xinepa

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change of Visual Analogue Scale (VAS) from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  It is a scale for the assessment of pain and it's based on a ten point scale, where 0 means no pain and 10 the greatest pain ever both at rest and during movements.

SECONDARY OUTCOMES:
Change of Semmes-Weinstein Monofilaments of light touch and pressure sensation test from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  Involves the use of five monofilaments of different colours that identify the levels of decrease in sensitivity, measurable, necessary for the evaluation of the perception of the surface touch.
Change of Boston Carpal Tunnel Questionnaire from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  It consists of two scales, the scale of the severity of symptoms (SSS) and functional status scale (FSS). The first includes the first 11 questions relating to: the intensity of pain during the day and night, lasting pain during the day, sleep, weakness, tingling sensation during the night and its frequency and abilities. Each question provides a metric scale ranging from 1 (absence of symptoms) to 5 (severe symptoms). The second scale includes the last eight questions concerning activities such as writing, buttoning clothes, hold a book while reading, hold up the phone, clean, carry bags, open the lid of a jar.
Change of the measurement of the grip strength trough the Jamar dynamometer from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  It consists of a manometer with a double scale to recorder static force in kilos and pounds and a handle with 5 different positions of increasing amplitude from 3.5 cm to 8.8 cm. The patient holds the dynamometer and performs a grip at maximum force. The final score originates from the average of three measurements taken for each position of the handle.
Change of the measurement of the pinch strength trough the Pinch Gauges dynamometer from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  It consists of a manometer with a double scale to recorder static force in kilos and libbre and two caliper levers with the tips away from each other of 2.2 cm/ 1.9 cm. Three types of pliers are evaluated: side, three tips, tip against tip. The patient holds the dynamometer and performs a grip at maximum force. The final score originates from the average of three measurements taken for each type of tongs.
Change of electroneurography from baseline to 12 months | baseline, 4 weeks, 12 weeks
  It allows the study of nerve of the median nerve (speed of motor-sentitive run and latency).

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Maria Saraceni, Study Director — Umberto I hospital, Sapienza University of Rome
Locations (1):
- Umberto I Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided